CLINICAL TRIAL: NCT00777907
Title: Complete Occlusion of Coilable Aneurysms
Acronym: COCOA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chestnut Medical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLP-0004
Record Dates: First submitted 2008-10-20; First posted 2008-10-22 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Intracranial Aneurysm
Keywords: neurovascular embolization; therapeutic embolization
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coil embolization (Active Comparator): Placement of bare platinum coils into the target aneurysm with balloon remodeling allowed. Stents are not allowed in this arm.
  Interventions: Device: Coil embolization
- Pipeline (Experimental): Placement of 1 or more Pipeline Embolization Device(s)(PED) into the parent artery at the target aneurysm.
  Interventions: Device: Pipeline Embolization Device (PED)

INTERVENTIONS:
Device: Pipeline Embolization Device (PED) — 1 or more PEDs placed in the parent artery of the affected aneurysm via endovascular approach.
  Other Names: Pipeline Embolization Device, PED
  Arms: Pipeline
Device: Coil embolization — Placement of bare platinum coils into the target aneurysm with balloon remodeling allowed.
  Arms: Coil embolization

SUMMARY:
To compare the safety and effectiveness of Pipeline Embolization Device to coil embolization for the treatment of coilable wide-necked intracranial aneurysms

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 75 years, inclusive
* Patient has a single target IA that:

  1. is located in the following regions of the internal carotid artery: i. Paraophthalmic (including paraclinoid, ophthalmic and hypophyseal segments) ii. Cavernous iii. Petrous
  2. is saccular
  3. has a parent vessel with diameter 2.5-5.0 mm
* If target IA has a neck >4 mm, at least 2 of 3 members of an independent expert committee (IEC) have confirmed that coil embolization with optional adjunctive techniques** has a very high likelihood of procedural success (i.e., coil placement and retention)
* Subject has provided written informed consent using the IRB-approved consent form
* Subject has the necessary mental capacity to participate and is willing and able to comply with protocol requirements

  * ** Adjunctive techniques include intravascular balloons ["balloon remodeling"], 3D coils, dual catheter techniques.

Exclusion Criteria:

* Target IA has BOTH neck >4 mm AND size (maximum fundus diameter) >10 mm
* More than one IA requires treatment in the next 6 months
* Subarachnoid hemorrhage in the past 60 days
* Any intracranial hemorrhage in the last 42 days
* Major surgery in the last 42 days
* Coils in place in the target IA
* Unstable neurologic deficit (i.e., any worsening of clinical condition in the last 30 days)
* Known irreversible bleeding disorder
* Platelet count < 100 x 103 cells/mm3 or known platelet dysfunction
* Inability to tolerate, documented evidence of adverse reaction or contraindication to study medications
* Prior stent placement at target site
* Contraindication to CT scan AND MRI
* Known allergy to contrast used in angiography that cannot be medically controlled
* Known severe allergy to platinum or cobalt/chromium alloys
* Relative contraindication to angiography (e.g., serum creatinine > 2.5 mg/dL)
* Woman of child-bearing potential who cannot provide a negative pregnancy test
* Evidence of active infection at the time of treatment
* Other known conditions of the heart, blood, brain or intracranial vessels that carry a high risk of neurologic events (e.g., severe heart failure, atrial fibrillation, known carotid stenosis)
* Current use of cocaine or other illicit substance
* Any comorbid disease or condition expected to compromise survival or ability to complete follow-up assessments to 180 days
* Extracranial stenosis greater than 50% in the carotid artery
* Intracranial stenosis greater than 50% in the treated vessel

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-10; Primary Completion 2014-11 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Effectiveness: Proportion of subjects whose target aneurysm shows complete occlusion on angiogram with <=50% stenosis of the parent artery. Safety: Proportion of subjects with ipsilateral major stroke or neurologic death. | 180 days

SECONDARY OUTCOMES:
Rate of complete target aneurysm occlusion | 1, 3 and 5 years
Incidence of ipsilateral major stroke | 180 days
Change in modified Rankin scale (MRS) | 180 days, 1, 3 and 5 years
Incidence of device-related adverse events | 180 days, 1, 3 and 5 years
Change from baseline in neurologic signs or symptoms related to the target aneurysm | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: David Fiorella, MD, PhD, Principal Investigator — Barrow Neurologic Institute
Locations (2):
- United States (2):
  - Barrow Neurological Institute, Phoenix, Arizona
  - SUNY Stony Brook, Stony Brook, New York